CLINICAL TRIAL: NCT03269786
Title: Laoboratory and Ultrasonographic Changes After Endoscopic Varisceal Treatment
Brief Title: Changes in Lab and Ultrasonography After Endoscopic Varisceal Treatment
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mahmoud Abdelhamed, principal investigator, Assiut University
Other Study IDs: laucaevt
Record Dates: First submitted 2017-08-27; First posted 2017-09-01 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Liver Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis | interventions — Liver Function Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- cirrhotic patients with esophagel varisces: Endoscopic band ligation or injection scelerotheraby will be done for all patients
  Interventions: Diagnostic Test: Liver function tests (ALT,AST,ALBUMIN,BILIRUBIN,INR,PC,CBC); Device: biannual ultrasonography

INTERVENTIONS:
Diagnostic Test: Liver function tests (ALT,AST,ALBUMIN,BILIRUBIN,INR,PC,CBC) — Liver function tests will be assessed after endoscopic varisceal treatment for 6 monthes
Device: biannual ultrasonography — portal vein diameter , portal vein velocity and flow direction, volume flow in portal vein , congetive index, spleen size.will be assessed after endoscopic varisceal treatment by using biannual ultrasonography for 6 monthes

SUMMARY:
laboratory and ultrasongraphicc changes after endoscopical varices treatment

ELIGIBILITY:
Inclusion Criteria:

* patients with liver cirrhosis and portal hyprtension with esophagel varisces

Exclusion Criteria:

* 1. Patients with heart failure or renal failure 2. patients with COPD 3. Patients with hepato cellular carcinoma and portal vein thrombosis 4. Pregnant

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: patients with liver cirrhosis and portal hyprtension with esophagel varisces
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-11-01 (Estimated); Primary Completion 2019-11-01 (Estimated); Study Completion 2019-11-01 (Estimated)

PRIMARY OUTCOMES:
Changes in liver function tests | 6 months
  Liver function tests (ALT, AST, bilirubin,Albumin,Cbc,Prothrombin time,INR ) level (expected to be lower after endoscopic varisceal treatment
  (ex
Ultrasonographic changes | 6 months
  { portal vein diameter , portal vein velocity and flow direction, volume flow in portal vein , congetive index, spleen size.(expected to be chnged after endoscopic varisceal treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No